CLINICAL TRIAL: NCT04830202
Title: Expanded Access to Telisotuzumab Vedotin
Status: Available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C20-503
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Non-Small Cell Lung Cancer (NSCLC); Telisotuzumab vedotin; ABBV-399; Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — telisotuzumab vedotin

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Telisotuzumab vedotin — Intravenous Infusion
  Other Names: ABBV-399

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to Telisotuzumab vedotin prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Exclusion Criteria:

* There are other suitable treatment options.
* The participant qualifies for ongoing clinical trials.

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie